CLINICAL TRIAL: NCT01221493
Title: EBUS Guided Cryo Biopsy of Solitary Pulmonary Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Felix JF Herth, Thoraxklinik, University of Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-320
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-03

CONDITIONS: Yield of Cryo Biopsy in Lung Cancer; Solitary Pulmonary Nodule
Keywords: solitary pulmonary nodules; transbronchial lung biopsy; endobronchial ultrasound
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryo biospy (Experimental)
  Interventions: Procedure: Cryo biopsy

INTERVENTIONS:
Procedure: Cryo biopsy — Cryoprobe, Erbe Company
  Other Names: Cryo biopsy probe 20416-032, ERBE company, Germany

SUMMARY:
To proof the feasibility and safety of EBUS guided transbronchial cryo biopsies in peripheral lung lesions

DETAILED DESCRIPTION:
Solitary pulmonary nodule are a diagnostic dilemma. Nowadays not only the basic tissue diagnosis is necessary, molecular signals are state of the art. Therefore more tissue is necessary. With a cryoprobe the amount of tissue is increased compared to the classical forceps biopsy.

Until now, the use of the cryoprobe ism´t show in peripheral lung tissue.

ELIGIBILITY:
Inclusion Criteria:

* solitary pulmonary nodule < 4 cm
* no endobronchial lesion
* indication for bronchoscopy

Exclusion Criteria:

* coagulopathy
* pulmonary hypertension
* pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 24 h after intervention
  Number of Participants with Adverse Events as a Measure of Safety Detailed analysis of number of Pneumothoraces and number of bleeding complication

SECONDARY OUTCOMES:
Efficacy | 48 h after intervention
  Diagnostic yield of the different biopsy techniques in establishing a specific diagnosis of the lesion

CONTACTS AND LOCATIONS:
Overall Officials: Felix JF Herth, MD, PhD, Principal Investigator — Thoraxklinik, Universityof Heidelberg
Locations (1):
- Department of Pneumology and Critical Care medicine, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Eberhardt R, Kahn N, Gompelmann D, Schumann M, Heussel CP, Herth FJ. LungPoint--a new approach to peripheral lesions. J Thorac Oncol. 2010 Oct;5(10):1559-63. doi: 10.1097/JTO.0b013e3181e8b308. PMID 20802352
- [Background] Eberhardt R, Gompelmann D, Herth FJ. Electromagnetic navigation in lung cancer: research update. Expert Rev Respir Med. 2009 Oct;3(5):469-73. doi: 10.1586/ers.09.36. PMID 20477337
- [Background] Eberhardt R, Morgan RK, Ernst A, Beyer T, Herth FJ. Comparison of suction catheter versus forceps biopsy for sampling of solitary pulmonary nodules guided by electromagnetic navigational bronchoscopy. Respiration. 2010;79(1):54-60. doi: 10.1159/000232394. Epub 2009 Jul 31. PMID 19648733
- [Background] Eberhardt R, Kahn N, Herth FJ. 'Heat and destroy': bronchoscopic-guided therapy of peripheral lung lesions. Respiration. 2010;79(4):265-73. doi: 10.1159/000284015. Epub 2010 Feb 10. PMID 20203535
- [Derived] Schuhmann M, Bostanci K, Bugalho A, Warth A, Schnabel PA, Herth FJ, Eberhardt R. Endobronchial ultrasound-guided cryobiopsies in peripheral pulmonary lesions: a feasibility study. Eur Respir J. 2014 Jan;43(1):233-9. doi: 10.1183/09031936.00011313. Epub 2013 Jul 30. PMID 23900983